CLINICAL TRIAL: NCT05984264
Title: Efficacy of Topical Lidocaine/Prilocaine in Pain Management in Pleurocentesis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Abd El-gayed Eid, Fellow, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBBAAS
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion | interventions — Lidocaine; Prilocaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pridocaine cream (Experimental): Pridocaine cream (lidocaine 2.5% and prilocaine 2.5%) will be applied at least 30 min before the pleurocentesis on the skin overlying the chosen aspiration site using ultrasound under occlusive dressing over a 5 × 5 cm area.
  Interventions: Drug: lidocaine 2.5% and prilocaine 2.5% cream in pain management before pleurocentesis.
- Standardized local lidocaine infiltration (Active Comparator): Anesthetize the skin over the insertion site with 1% lidocaine using the 5 ml syringe with a 25 or 27-gauge needle. Next, anesthetize the superior surface of the rib and the pleura. The needle is inserted over the top of the rib (superior margin) to avoid the intercostal nerves and blood vessels that run on the underside of the rib (the intercostal nerve and the blood supply are located near the inferior margin). As the needle is inserted, aspirate back on the syringe to check for pleural fluid. Once fluid returns, note the depth of the needle and mark it with a hemostat. This gives an approximate depth for the insertion of the thoracentesis needle. Remove the anesthetizing needle.
  Interventions: Drug: lidocaine 2.5% and prilocaine 2.5% cream in pain management before pleurocentesis.

INTERVENTIONS:
Drug: lidocaine 2.5% and prilocaine 2.5% cream in pain management before pleurocentesis. — Pridocaine cream (lidocaine 2.5% and prilocaine 2.5%) will be applied at least 30 min before the pleurocentesis on the skin overlying the chosen aspiration site using ultrasound under occlusive dressing over a 5 × 5 cm area. The time interval between topical Pridocaine cream (lidocaine 2.5% and prilocaine 2.5%) application and pleural aspiration will be 30 min, and 45 min.
  Other Names: Pridocaine cream in pain management before pleurocentesis.

SUMMARY:
The research aims to compare the efficacy of topical Pridocaine cream (lidocaine 2.5% and prilocaine 2.5%) and the standardized local lidocaine infiltration in pain management before pleurocentesis.

DETAILED DESCRIPTION:
Acute pain management is a core ethical concept in medical practice. During pleurocentesis, the standardized pain management is with 1% lidocaine with a 25 gauge needle for skin and a smaller gauge needle for deeper tissue. As the anesthetic injection is painful in and of itself, during these two procedures, pain management can sometimes fall short due to a lack of education and incorrect personal opinions. One example is "one needle insertion can cause less pain than two-needle insertions". Therefore, it is essential to find an alternative method that is painless and reduces procedural pain, which does not require expertise to administer. This is particularly important in centers with a high volume of patients and a lack of expert medical staff.

Another option for administering a local anesthesia is using a topical anesthetic. Generally, these are easily applied, tolerated better by patients, and have minimal systemic absorption resulting in fewer side effects6. A topical anesthetic can be a substitute for infiltrative lidocaine (IL) if it can be effective in reducing pain. Lidocaine-prilocaine cream (LPC) is an example of a topical anesthetic, which was introduced in 1980 for dermabrasion and minor surgery.

Previous research findings had noted the efficacy of LPC compared to IL in trans-radial catheterization, perineal tears following vaginal delivery, and some pediatric procedures like lumbar punctures and venipunctures. Additionally, LPC can be substituted for infiltrative prilocaine in pediatric femoral catheterization.

Hanieh Halili et al, found a significant difference between the LPC and IL groups in terms of patient pain or satisfaction levels, but their study was on a small sample size and they recommended further studies.

ELIGIBILITY:
Inclusion Criteria:

* All Patients will be prepared for pleurocentesis.

Exclusion Criteria:

1. Patients with a known history of sensitivity to local anesthetics of the amide type or to any other component of the product.
2. Patients treated with class III anti-arrhythmic drugs (e.g., amiodarone, bretylium, sotalol, dofetilide).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The severity of pain will be assessed using the visual analogue scale (VAS). | one day
  The severity of pain will be assessed using the visual analogue scale (VAS). The VAS consists of a 10cm line, with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could be'). Ask the patient to rate their current level of pain by placing a mark on the line. Use a ruler to measure the distance in centimeters from the 'no pain marker' (or zero) to the current pain mark. This provides a pain intensity score out of 10; for example, 6 out of 10 (or 6/10).

CONTACTS AND LOCATIONS:
Overall Officials: Safaa A Eid, MD, Principal Investigator — Assiut University
Locations (1):
- Assuit University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Akbar N, Teo SP, Artini Hj-Abdul-Rahman HN, Hj-Husaini HA, Venkatasalu MR. Barriers and Solutions for Improving Pain Management Practices in Acute Hospital Settings: Perspectives of Healthcare Practitioners for a Pain-Free Hospital Initiative. Ann Geriatr Med Res. 2019 Dec;23(4):190-196. doi: 10.4235/agmr.19.0037. Epub 2019 Dec 23. PMID 32743311
- [Background] Patel BK, Wendlandt BN, Wolfe KS, Patel SB, Doman ER, Pohlman AS, Hall JB, Kress JP. Comparison of Two Lidocaine Administration Techniques on Perceived Pain From Bedside Procedures: A Randomized Clinical Trial. Chest. 2018 Oct;154(4):773-780. doi: 10.1016/j.chest.2018.04.018. Epub 2018 Apr 24. PMID 29698720
- [Background] Story M. One Needle is Better Than Two: The Philosophy Surrounding Use of Local Anesthesia in Northern India. J Pain Palliat Care Pharmacother. 2017 Jun;31(2):162-164. doi: 10.1080/15360288.2017.1298687. Epub 2017 Mar 27. PMID 28346035
- [Background] Halili H, Azizkhani R, Tavakoli Garmaseh S, Jafarpisheh MS, Heydari F, Masoumi B, Maghami Mehr A. Comparing the Effect of Lidocaine-Prilocaine Cream and Infiltrative Lidocaine on Overall Pain Perception During Thoracentesis and Abdominocentesis: A Randomized Clinical Trial. Anesth Pain Med. 2020 Nov 18;11(1):e106275. doi: 10.5812/aapm.106275. eCollection 2021 Feb. PMID 34249663
- [Background] You P, Yuan R, Chen C. Design and evaluation of lidocaine- and prilocaine-coloaded nanoparticulate drug delivery systems for topical anesthetic analgesic therapy: a comparison between solid lipid nanoparticles and nanostructured lipid carriers. Drug Des Devel Ther. 2017 Sep 18;11:2743-2752. doi: 10.2147/DDDT.S141031. eCollection 2017. PMID 29075099
- [Background] Latsios G, Toutouzas K, Antonopoulos AS, Melidi E, Synetos A, Vogiatzi G, Stasinopoulou A, Tsioufis K, Tsiamis E, Tousoulis D. Anesthetic ointment only (lidocaine/prilocaine) instead of injectable local lidocaine in trans-radial catheterization: A viable no-needle alternative. J Interv Cardiol. 2017 Aug;30(4):382-386. doi: 10.1111/joic.12399. Epub 2017 Jun 26. PMID 28653424
- [Background] Abbas AM, Abdel Hafiz HA, Abdelhafez AM, Michael A, Ismail AM. Topical lidocaine-prilocaine cream versus lidocaine infiltration for pain relief during repair of perineal tears after vaginal delivery: randomized clinical trial. J Matern Fetal Neonatal Med. 2019 Jul;32(13):2182-2187. doi: 10.1080/14767058.2018.1428304. Epub 2018 Jan 31. PMID 29334290
- [Background] Cruickshank A, Qeadan F, Kuttesch JF, Agarwal HS. Eutectic mixture of lidocaine and prilocaine versus 1% lidocaine injection for lumbar punctures in pediatric oncology patients. Pediatr Blood Cancer. 2019 Nov;66(11):e27957. doi: 10.1002/pbc.27957. Epub 2019 Aug 18. PMID 31423750
- [Background] Pirat A, Karaaslan P, Candan S, Zeyneloglu P, Varan B, Tokel K, Torgay A, Arslan G. Topical EMLA cream versus prilocaine infiltration for pediatric cardiac catheterization. J Cardiothorac Vasc Anesth. 2005 Oct;19(5):642-5. doi: 10.1053/j.jvca.2004.10.007. PMID 16202900
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Qureshi AI, Saleem MA, Naseem N, Aytac E, Akpinar CK, Wallery SS. Effectiveness of Topical Lidocaine-Prilocaine Cream for Pain Control During Femoral Artery Catheterization in Adult Patients: A Prospective Study. J Vasc Interv Neurol. 2018 Jun;10(1):60-64. PMID 29922408
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- [Background] Tihan D, Totoz T, Tokocin M, Ercan G, Koc Calikoglu T, Vartanoglu T, Celebi F, Dandin O, Kafa IM. Efficacy of laparoscopic transversus abdominis plane block for elective laparoscopic cholecystectomy in elderly patients. Bosn J Basic Med Sci. 2016 Jan 14;16(2):139-44. doi: 10.17305/bjbms.2016.841. PMID 26773187